CLINICAL TRIAL: NCT00002900
Title: A STUDY OF THE LATE CARDIAC EFFECTS OF TWO DIFFERENT ADJUVANT CHEMOTHERAPY REGIMENTS IN WOMEN WITH NODE NEGATIVE BREAST CANCER TREATED ON SWOG-8897
Brief Title: SWOG-9342 Chemotherapy in Treating Women Enrolled in the SWOG-8897 Clinical Trial
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000065237; U10CA032102 (NIH); SWOG-9342
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer; Cardiac Toxicity
Keywords: stage I breast cancer; stage II breast cancer; ductal breast carcinoma; cardiac toxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Carcinoma, Ductal, Breast

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This clinical trial is studying the effect of chemotherapy on heart function in treating women who have breast cancer with negative axillary lymph nodes and who are undergoing treatment on the SWOG-8897 clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the frequency of subclinical congestive heart failure by measuring resting MUGA at 5-8 and 10-11 years after randomization in women receiving adjuvant chemotherapy with cyclophosphamide, methotrexate, and fluorouracil or cyclophosphamide, doxorubicin, and fluorouracil on protocol SWOG-8897.
* Estimate the frequency of late cardiac effects (congestive heart failure, cardiac ischemic events, and clinical symptoms) in these patients treated with these regimens.
* Monitor prospectively the incidence of annual cardiac events between the fifth and tenth year after randomization of these patients to these regimens.

OUTLINE: This is a multicenter study.

The treating physician completes patient cardiovascular and routine history and physical examination questionnaires at baseline and yearly. Patients undergo resting MUGA scans at 5-8 and 10-11 years after registration on protocol SWOG-8897. The first scan must be performed within 3 months prior to enrollment or within 1 month after registration on the current study, and the second scan must be done in the tenth year of follow-up and within 3 months prior to enrollment or 1 month from the anniversary of registration on the current study.

PROJECTED ACCRUAL: A total of 420 patients will be accrued for this study. After initial accrual is completed, approximately 50 additional patients will be accrued at 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women registered on Arm I, II, III, or IV of protocol SWOG-8897 who have completed at least 1 course of assigned chemotherapy

  * Completion of tamoxifen therapy not required
  * Registration to current study required between 5.25-8 years or 10-11 years after randomization to protocol SWOG-8897
* Patients must be diagnosed disease-free with no prior recurrence after registration on protocol SWOG-8897
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Pre- and postmenopausal

Performance status:

* Not specified

Life Expectancy:

* At least 5 years

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Pregnant or nursing women not eligible for nuclear medicine (MUGA) portion of study
* Fertile patients must use effective contraception during and for 1 month after MUGA

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior chemotherapy for second primary malignancy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for second primary malignancy

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven invasive adenocarcinoma of the breast with negative axillary lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 1997-02; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Ganz, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (105):
- United States (105):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Danville Radiation Therapy Center, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Ganz PA, Green SJ, Hutchins L, et al.: Late cardiac effects of adjuvant CMF vs CAF in women with node negative breast cancer treated on SWOG 8897: initial results from SWOG 9342. [Abstract] Breast Cancer Res Treat 76 (Suppl 1): A-10, 2002.